CLINICAL TRIAL: NCT06176560
Title: A Randomised, Double-blind, Double-dummy, Multicentre, Phase III, Non Inferiority Trial of an Oral Mesalazine Formulation in Patients With Active Mild to Moderate Ulcerative Colitis for the Induction of Remission.
Brief Title: Phase III Multicentre Trial of Oral Mesalazine in Patients With Mild to Moderate Ulcerative Colitis.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CGRA-0121/ES
Record Dates: First submitted 2023-12-04; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesalazine Experimental (Experimental): Mesalazine oral formulation
  Interventions: Drug: Mesalazine
- Mesalazine Comparator (Active Comparator): Mesalazine oral formulation
  Interventions: Drug: Mesalazine

INTERVENTIONS:
Drug: Mesalazine — Oral Formulation

SUMMARY:
A randomised, double-blind, double-dummy, multicentre, phase III, non inferiority trial of an oral mesalazine formulation in patients with active mild to moderate ulcerative colitis for the induction of remission.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age.
2. Provide written informed consent.
3. Be willing and able to follow all instructions, undergo all assessments, complete the electronic diary and attend all trial visits.
4. Have UC symptoms with UC diagnosis established by clinical, histological and endoscopic evidence.
5. Have active, mild to moderate UC at the time of screening.
6. Have a recent colonoscopy documenting the degree and extent of mucosal inflammation; otherwise, a colonoscopy must be performed during the screening period.
7. Be able and willing to avoid all disallowed medications for the appropriate washout period before randomisation and during the rest trial.
8. For females of childbearing potential only: willing to perform pregnancy tests, must agree to use effective methods of birth control throughout the trial until the trial ends. Effective methods of birth control include: combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (provided that partner is the sole sexual partner of the clinical trial patient and has documentation of azoospermia) or sexual abstinence (if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial treatment). The investigator is responsible for determining whether the patient has adequate birth control for trial participation.
9. For males with female partners of childbearing potential: acceptance to use birth control methods (condom with or without spermicide, or effective methods of birth control of female partner) throughout the trial duration and until 2.5 months after last intake of IMP. Vasectomy or sexual abstinence (if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial treatment) are also acceptable methods. The investigator is responsible for determining whether the patient has adequate birth control for trial participation.

Exclusion Criteria:

1. Have known contraindications or sensitivities to the use of the IMPs or any of its components.
2. History of difficulty in swallowing.
3. Be pregnant, planning a pregnancy or breastfeeding.
4. Have severe UC.
5. Have a history of colonic resection (excluding appendectomy).
6. Present moderate to severe renal disorder.
7. Present moderate to severe hepatic disorder.
8. Have a gastrointestinal disease that in the opinion of the investigator, would have interfered with the patient's participation in this study. Including but not limited to: Crohn's disease, other forms of colitis, coeliac disease, malabsorption syndromes, present or past colorectal cancer, gastric or duodenal ulcer.
9. Have ulcerative proctitis (restricted to rectum).
10. Suspected or documented infectious enterocolitis.
11. Have previous or current treatment with thiopurines, calcineurin inhibitors, methotrexate, JAK inhibitors and/or biologics.
12. Patients who previously were refractory to treatment with oral or rectal mesalazine.
13. Have a history of or current diagnosis of severe or uncontrolled pulmonary disease, myocarditis or pericarditis.
14. Severe or uncontrolled asthma, that in the opinion of the investigator, would compromise the patient safety.
15. Have a history of or current diagnosis of haemorrhagic diathesis.
16. Have an active malignancy or treatment with antineoplastic agents during the last 5 years. Patients with a history of cancer other than colorectal cancer and at least 5 years of uneventful follow-up and no signs of recurrence may be eligible according to the investigator's decision.
17. Have participated in another clinical trial in which an investigational drug (including investigational vaccines) or invasive investigational medical device has been taken within the past 90 days (or five half-lives of IMP whichever is longer) prior to Visit 1, or simultaneous participation in another clinical trial.
18. Have any condition that, in the opinion of the investigator, may jeopardise the clinical trial conduct according to the protocol.
19. Be an employee of the investigator or clinical trial unit, with direct involvement in the proposed trial or other studies under the direction of that investigator or clinical trial unit, as well as family members of the employees or the principal investigator.
20. Patients unable to understand the informed consent or having a high probability of non-compliance with the trial procedures.
21. Be a person committed to an institution by virtue of an order issued either by judicial or other authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To assess the percentage of patients with clinical remission [Mayo Modified Score (MMS) ≤ 2] and Endoscopic remission [Mayo Endoscopic Score (MES) ≤ 1] after 8 weeks of treatment. | 8 weeks

SECONDARY OUTCOMES:
To assess the percentage of patients achieving symptomatic remission using Modified Mayo Score. | 8 weeks
  Symptomatic remission defined by Modified Mayo Score (MMS)
To assess the percentage of patients achieving endoscopic remission using Mayo Endoscopic Score. | 8 weeks
  Endoscopic Remission defined by Mayo Endoscopic Score (MES)
To assess the percentage of patients achieving overall response using Mayo Modified Score | 8 weeks
  Reduction in Mayo Modified Score (MMS) from baseline with a decrease of rectal bleeding subscore.
To evaluate changes in the symptomatic assessments using Mayo Modified Score. | 8 weeks
  Mayo modified score: stool frequency and rectal bleeding.
To evaluate changes in the endoscopic score using Mayo Endoscopic Score. | 8 weeks
  Mayo Endoscopic Score
To assess the histological remission using Robarts Histopathology Index | 8 weeks
  Histologic Remission defined by Robarts Histopathology Index (RHI).
To assess the percentage of patients achieving overall remission | 8 weeks
  All modified Mayo subscores = 0
To assess patients' quality of life | 8 weeks
  Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
To evaluate change in faecal calprotectin. | 8 weeks
  Stool sample for faecal calprotectin analysis
To evaluate the safety and tolerability by incidence of AEs. | 8 weeks
To evaluate the safety and tolerability by clinically significant laboratory results. | 8 weeks
  Number of patients with clinically significant results at Week 8 in haematological, biochemistry and urinalysis parameters.
To evaluate the safety and tolerability by assessing clinically significant vital signs results. | 8 weeks
  Number of patients with clinically significant changes in vital signs parameters (blood pressure, heart rate and body temperature) from baseline to Week 8.
To evaluate the safety and tolerability by clinically significant physical examination findings. | 8 weeks
  Number of patients with clinically significant findings in physical examination (heart, lungs, abdomen) from baseline to Week 8.
To evaluate the safety and tolerability considering the percentage of patients withdrawn from the trial due to safety concerns. | 8 weeks

IPD SHARING:
Plan to Share IPD: No